CLINICAL TRIAL: NCT03332290
Title: Post Traumatic Stress Disorder (PTSD): Benefits of Diving Practice on Patient Quality of Life
Brief Title: Diving for Post Traumatic Stress Disorder (PTSD)
Acronym: Dive-Hope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marion Trousselard (Other Government)
Responsible Party: Sponsor-Investigator, Marion Trousselard, principal investigator, Institut de Recherche Biomedicale des Armees
Organization: Institut de Recherche Biomedicale des Armees (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-002436-16
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-01

CONDITIONS: Ptsd
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: randomized opened clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sport training (Active Comparator): training course lasting 10 days. It included 10 days of multisports practice once (2h) per day.
  Interventions: Behavioral: sport practice
- diving (Experimental): diving course lasting 10 days. It included 10 days of diving once (2h) per day. Diving will be carried out using air at a maximum depth of 30-meters
  Interventions: Behavioral: sport practice

INTERVENTIONS:
Behavioral: sport practice — the intervention was a training course lasting 10 days. It included 10 days of sports practice. For divers, diving was carried out using air at a maximum depth of 40-meters, with a maximum of one dives a day. For the multisport group (the non-divers), the course included kayaking, mountain climbing or hiking with a maximum of two activities a day.

SUMMARY:
within the components of Scuba diving there are similarities with meditation and mindfulness techniques. PTSD and emotion dysregulation are known to be involved by meditation training This study evaluates the benefits of scuba diving on quality of life and mindful functioning comparing the benefits of diving training using a clinical trial protocol

ELIGIBILITY:
Inclusion Criteria:

* ptsd

Exclusion Criteria:

* mindfulness practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
quality of life (Mental Health Continuum-Short Form (MHC-SF)) | changes from baseline (after the course minus baseline), (1month after the course minus baseline) and (3months after the course minus baseline)
  four times (baseline, after the course, 1month after the course and 3months after the course)

SECONDARY OUTCOMES:
post-traumatic checklist scale; a 20-item self-report scale assessing the 20 DSM-5 symptoms of PTSD with a symptom severity from 0 to 80 and a cut-point score of 33. | changes from baseline (after the course minus baseline), (1month after the course minus baseline) and (3months after the course minus baseline
  four times (baseline, after the course, 1month after the course and 3months after the course)
heart rate variability on morning | changes from baseline (after the course minus baseline), (1month after the course minus baseline) and (3months after the course minus baseline
  four times (baseline, after the course, one month after the course and 3 months after the course)

CONTACTS AND LOCATIONS:
Locations (1):
- Marion Trousselard, Brétigny-sur-Orge, Not in US/Canada, France

IPD SHARING:
Plan to Share IPD: Undecided